CLINICAL TRIAL: NCT04237493
Title: Effect of Dosage Reduction of Glucose-Lowering Multidrug Regimens on the Incidence of Acute Glycemic Complications in People With Type 2 Diabetes Who Fast During Ramadan: An Open-Label, Parallel-Group, Randomized, Controlled Trial
Brief Title: Dosage Reduction and Acute Glycemic Complications in People With Type 2 Diabetes Who Fast During Ramadan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Ayman A. Zayed, MD, Professor of Medicine, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 671201612222
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Fasting; Hypoglycemic Agents; Hypoglycemia; Hyperglycemia; Diabetic Ketoacidosis; Hyperglycemic Hyperosmolar Nonketotic Coma; Metformin; Glimepiride; Vildagliptin; Insulin Glargine; Insulin, Regular, Human
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fasting; Hypoglycemia; Hyperglycemia; Diabetic Ketoacidosis; Hyperglycemic Hyperosmolar Nonketotic Coma; Insulin Resistance | interventions — Metformin; glimepiride; Vildagliptin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-dosage therapy (Experimental)
  Interventions: Drug: Metformin and Glimepiride (Low Dosage); Drug: Metformin and Vildagliptin (Low Dosage); Drug: Metformin and Insulin Glargine U100 (Low Dosage); Drug: Metformin, Insulin Glargine U100, and Human Regular Insulin (Low Dosage)
- Regular-dosage therapy (Active Comparator)
  Interventions: Drug: Metformin and Glimepiride (Regular Dosage); Drug: Metformin and Vildagliptin (Regular Dosage); Drug: Metformin and Insulin Glargine U100 (Regular Dosage); Drug: Metformin, Insulin Glargine U100, and Human Regular Insulin (Regular Dosage)

INTERVENTIONS:
Drug: Metformin and Glimepiride (Low Dosage) — * Metformin (PO; 850 mg; BID [with Ifṭār and with Suḥūr])
  * Glimepiride (PO; 1.5 or 3 mg [75% of the pre-Ramadan dose]; OD [with Ifṭār])
  Arms: Low-dosage therapy
Drug: Metformin and Vildagliptin (Low Dosage) — * Metformin (PO; 850 mg; BID [with Ifṭār and with Suḥūr])
  * Vildagliptin (PO; 50 mg; OD [with Ifṭār])
  Arms: Low-dosage therapy
Drug: Metformin and Insulin Glargine U100 (Low Dosage) — * Metformin (PO; 850 mg; BID [with Ifṭār and with Suḥūr])
  * Insulin Glargine U100 (SC; 9-33 units [75% of the pre-Ramadan dose]; OD [at 10 P.M.])
  Arms: Low-dosage therapy
Drug: Metformin, Insulin Glargine U100, and Human Regular Insulin (Low Dosage) — * Metformin (PO; 850 mg; BID [with Ifṭār and with Suḥūr])
  * Insulin Glargine U100 (SC; 6-39 units (75% of the pre-Ramadan dose); OD [at 10 P.M.])
  * Human Regular Insulin (SC; 15-33 units before Ifṭār and 6-18 units before Suḥūr [75% of the pre-Ramadan doses])
  Arms: Low-dosage therapy
Drug: Metformin and Glimepiride (Regular Dosage) — * Metformin (PO; 850 mg; BID [with Ifṭār and with Suḥūr])
  * Glimepiride (PO; 2 or 4 mg [100% of the pre-Ramadan dose]; OD [with Ifṭār])
  Arms: Regular-dosage therapy
Drug: Metformin and Vildagliptin (Regular Dosage) — * Metformin (PO; 850 mg; BID [with Ifṭār and with Suḥūr])
  * Vildagliptin (PO; 50 mg; BID [with Ifṭār and with Suḥūr]])
  Arms: Regular-dosage therapy
Drug: Metformin and Insulin Glargine U100 (Regular Dosage) — * Metformin (PO; 850 mg; BID [with Ifṭār and with Suḥūr])
  * Insulin Glargine U100 (SC; 11-44 units [100% of the pre-Ramadan dose]; OD [at 10 P.M.])
  Arms: Regular-dosage therapy
Drug: Metformin, Insulin Glargine U100, and Human Regular Insulin (Regular Dosage) — * Metformin (PO; 850 mg; BID [with Ifṭār and with Suḥūr])
  * Insulin Glargine U100 (SC; 8-52 units (100% of the pre-Ramadan dose); OD [at 10 P.M.])
  * Human Regular Insulin (SC; 12-40 units before Ifṭār and 7-28 units before Suḥūr [100% of the pre-Ramadan doses])
  Arms: Regular-dosage therapy

SUMMARY:
Every lunar year, during the month of Ramadan, Muslims abstain from food and drink between dawn and nightfall. People with type 2 diabetes who fast during Ramadan are at an increased risk of acute glycemic complications. Our aim is to investigate the effect of dosage reduction of four glucose-lowering multidrug regimens on the incidence of acute glycemic complications in people with type 2 diabetes who fast during Ramadan.

ELIGIBILITY:
Inclusion Criteria:

* Prospective participant is a returning patient with type 2 diabetes;
* Prospective participant expressed an intention to fast during Ramadan;
* Prospective participant has been compliant with one of four glucose-lowering multidrug regimens for at least the past three months.

Exclusion Criteria:

* Prospective participant is a pregnant, postpartum, breastfeeding, or eumenorrheic woman;
* Prospective participant has experienced diabetic ketoacidosis or hyperosmolar hyperglycemic state within three months;
* Prospective participant has received niacin or corticosteroids within one month; and,
* Prospective participant has any history of recurrent hypoglycemia, hypoglycemia unawareness, chronic renal insufficiency (stages IV or V), liver cirrhosis, uncontrolled epilepsy, depressive disorder, bipolar disorder, psychotic disorder, or cognitive dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 687 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia | 29 days of Ramadan
  Incidence of hypoglycemia
Hyperglycemia | 29 days of Ramadan
  Incidence of hyperglycemia

SECONDARY OUTCOMES:
Diabetic ketoacidosis | 29 days of Ramadan
  Incidence of diabetic ketoacidosis
Hyperosmolar hyperglycemic state | 29 days of Ramadan
  Incidence of hyperosmolar hyperglycemic state

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A. Zayed, MD, Principal Investigator — The University of Jordan School of Medicine
Locations (1):
- Jordan University Hospital, Amman, Amman Governorate, Jordan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zaghlol LY, Beirat AF, Amarin JZ, Hassoun Al Najar AM, Hasan YY, Qtaishat A, Tierney ME, Zaghlol RY, Zayed AA. Effect of Dosage Reduction of Hypoglycemic Multidrug Regimens on the Incidences of Acute Glycemic Complications in People With Type 2 Diabetes Who Fast During Ramadan: A Randomized Controlled Trial. Front Endocrinol (Lausanne). 2021 Jul 7;12:613826. doi: 10.3389/fendo.2021.613826. eCollection 2021. PMID 34305809